CLINICAL TRIAL: NCT02642224
Title: Trauma Services Intervention to Prevent Violence
Acronym: TSI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Collaborators: The Pittsburgh Foundation (Other); Hillman Foundation (Unknown); RK Mellon Foundation (Unknown)
Responsible Party: Principal Investigator, Steven M. Albert, Professor and Chair, Principal Investigator, University of Pittsburgh
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: UN2013-67786
Record Dates: First submitted 2013-12-27; First posted 2015-12-30 (Estimated); Last update posted 2018-07-02 (Actual); Status verified 2018-06

CONDITIONS: Skin Injury Due to Violence; Gunshot Wound, Contact
Keywords: Violence; firearm; guns; homicide; trauma; injury
MeSH Terms: conditions — Wounds, Gunshot; Wounds and Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Social work intervention (Experimental): The National Network of Hospital Violence Intervention (NNHVI) suggests that intervening when gunshot victims are receiving treatment in hospital trauma services may be effective in linking high-risk individuals to appropriate case management services, and that this service linkage may lower the risk of further violence. Our adaptation of the NNHVI model will focus on the social networks of gunshot victims as well as the victims themselves. Intervention efforts will range from job training and mentoring to relocation to different communities.
  Interventions: Behavioral: Social Work Case Management

INTERVENTIONS:
Behavioral: Social Work Case Management — The National Network of Hospital Violence Intervention (NNHVI) suggests that intervening when gunshot victims are receiving treatment in hospital trauma services may be effective in linking high-risk individuals to appropriate case management services, and that this service linkage may lower the risk of further violence. Our adaptation of the NNHVI model will focus on the social networks of gunshot victims as well as the victims themselves. Intervention efforts will range from job training and mentoring to relocation to different communities.

SUMMARY:
Primary outcome: Research participants and their network contacts will be followed over 6 months to assess whether a social work case management protocol results in reduction of trauma services recidivism and criminal violence arrests.

DETAILED DESCRIPTION:
Allegheny County, PA continues to suffer between 100-120 homicides each year, with perhaps 2-3 times as many gunshot injuries that require hospitalization. Firearm homicides overwhelmingly affect African American men aged 15-35. Building on prior efforts in violence prevention, the investigators propose to launch a hospital trauma service intervention that will take advantage of a "teachable moment" in the emergency room. All four hospitals providing Level I Trauma services in Allegheny County have agreed to host the program, an evidence-based effort developed by the National Network of Hospital Violence Intervention (NNHVI). Adaptation of the NNHVI model will focus on the social networks of gunshot victims as well as the victims themselves. Intervention efforts will range from job training and mentoring to relocation to different communities. The investigators will offer the opportunity to participate in the research and receive the intervention to all gunshot victims identified in county Level I trauma services. Participants in the research protocol will be asked to recruit their high-risk social network members for the intervention.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18+
2. Gunshot victim treated and discharged from Level I trauma facility; or member of social network of gunshot victim who may be high risk of firearm violence -

Exclusion Criteria:

1. Gunshot wound because of suicide attempt
2. Gunshot wound because of non-violent episode (e.g., hunting accident)
3. Unable to participate in research interview because of cognitive deficit
4. Planning to leave community as result of shooting
5. Discharged from trauma service to prison
6. Unable to provide informed consent -

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 111 (Actual)
Dates: Start 2014-05; Primary Completion 2018-05 (Actual); Study Completion 2018-05 (Actual)

PRIMARY OUTCOMES:
Trauma services recidivism | 6 months
  Readmission to hospital trauma service because of firearm injury
Arrest for violent crime | 6 months
  Arrests involving criminal violence noted in DA docket

SECONDARY OUTCOMES:
Social work case management goals | 6 months
  Educational program enrollment, job training, receipt of drug and alcohol treatment, trauma counseling

CONTACTS AND LOCATIONS:
Overall Officials: Steven M Albert, PhD, Principal Investigator — University of Pittsburgh
Locations (1):
- University of Pittsburgh, Graduate School of Public Health, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes
Data will be archived and made available to qualified investigators